CLINICAL TRIAL: NCT04503798
Title: Rehabilitation of Executive Dysfunction in Nonamnestic MCI Using Online Goal Management Training®
Brief Title: Online Cognitive Rehabilitation of Executive Dysfunction in Nonamnestic MCI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Baycrest (Other)
Collaborators: Centre for Aging and Brain Health Innovation (Other)
Responsible Party: Principal Investigator, Brian Levine, Senior Scientist, Baycrest
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: #08-53
Record Dates: First submitted 2020-08-05; First posted 2020-08-07 (Actual); Last update posted 2020-08-07 (Actual); Status verified 2020-08

CONDITIONS: Nonamnestic Mild Cognitive Impairment; Cognitive Dysfunction; Cognitive Disorder; Neurocognitive Disorders; Mental Disorder; Cognitive Impairment, Mild
Keywords: nonamnestic MCI; executive functions; online cognitive intervention; online cognitive rehabilitation
MeSH Terms: conditions — Cognitive Dysfunction; Neurocognitive Disorders; Mental Disorders

STUDY DESIGN:
Intervention Model Description: Participants are screened, undergo a battery of tests at pre-test, and then are randomly assigned to one of two conditions: online GMT intervention or treatment-as-usual control group. After the intervention, the participants take the same test battery and complete it once more at 6 week follow-up.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The study personnel who conduct screening and send pre/post-test surveys to participants are all blinded.
  Randomizer is blinded to all participant pre-test outcomes. Care providers know what their participants are doing, but not aware of the full study design, including details of the other conditions or outcome test characteristics.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Online Goal Management Training (GMT) (Experimental): The online version of GMT with a therapist on the back-end monitoring progress and giving feedback throughout the program. Online GMT takes 5-9 weeks (self-paced) to complete 9 modules involving instructional video with interactive content, practice of cognitive strategies through games, and between-module exercises.
  Interventions: Behavioral: Online Goal Management Training
- Treatment-as-usual control group (No Intervention): Participants randomized to this arm will receive no additional information or access to the intervention program. They will continue to receive treatment-as-usual from their care providers.

INTERVENTIONS:
Behavioral: Online Goal Management Training — Pre-recorded videos and games combine psycho-education, targeted skills training, and mindfulness practice to teach a system where participants can take control of their attention and cognitive faculties.
  Other Names: GMT
  Arms: Online Goal Management Training (GMT)

SUMMARY:
Nonamnestic mild cognitive impairment (naMCI) is a prodromal state characterized by deficits in executive functioning, a collection of higher-order abilities involved in organization, planning, inhibition, and complex reasoning. Research shows that individuals with naMCI have an increased risk of developing non-Alzheimer's dementia such as frontotemporal dementia and dementia with Lewy bodies, which pose substantial personal and societal costs. Accordingly, interventions that can successfully slow down or reverse the course of naMCI are needed.

Goal Management Training (GMT) is a cognitive rehabilitation platform that has been studied extensively, applied clinically, and manualized into kits for clinicians (Levine et al., 2000; Levine et al., 2007; Levine et al., 2011; Stamenova & Levine, 2019). The purpose of GMT is to train individuals to periodically "STOP" what they are doing, attend to task goals, evaluate their performance, and monitor or check outcomes as they proceed. Recently, an online version of GMT has been developed and validated in order to circumvent barriers to attending in-person sessions.

The purpose of the current study is to determine if the online version of GMT is effective at improving self-reported executive dysfunction in individuals diagnosed with naMCI against a control group that is receiving treatment-as-usual from their care provider. It is hypothesized that, compared to the control group, individuals receiving GMT will report a decrease in executive function deficits.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of nonamnestic mild cognitive impairment
* Available to participate in all testing and intervention sessions
* Access to a computer
* Computer familiarity
* Normal or corrected-to-normal vision and hearing

Exclusion Criteria:

* Diagnosis of amnestic mild cognitive impairment or dementia
* Moderate to severe affective impairment defined by score above cut-off for depression on the Patient Health Questionnaire-9 (PHQ-9; Kroenke et al., 2001)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-08-20 (Estimated); Primary Completion 2021-10-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in dysexecutive functioning - participants' report | Pre-intervention; Immediately post-intervention; 6 weeks post-intervention
  Dysexecutive Functioning Index (DEX; Burgess et al., 1996) questionnaire measures self-reported deficits in executive functions, and is composed of one scale with scores ranging from 0-80, where higher scores indicate greater executive deficit.
Change in cognitive failures | Pre-intervention; Immediately post-intervention; 6 weeks post-intervention
  Cognitive Failures Questionnaire (CFQ; Broadbent et al., 1992) measures self-reported failures in perception, memory, and motor function. It contains a single scale with scores ranging from 0-100, where higher scores indicate greater degree of impairment.
Change in dysexecutive functioning - carers' report | Pre-intervention; Immediately post-intervention; 6 weeks post-intervention
  Dysexecutive Functioning Index (DEX; Burgess et al., 1996) questionnaire completed by participants carers'.

SECONDARY OUTCOMES:
Change in Cambridge Brain Sciences online cognitive assessment | Pre-intervention; Immediately post-intervention; 6 weeks post-intervention
  Battery of online tasks that assess aspects of memory and reasoning (Hampshire et al., 2012).
Change in associative memory | Pre-intervention; Immediately post-intervention; 6 weeks post-intervention
  Face-name task associative memory score (Troyer et al., 2012).

CONTACTS AND LOCATIONS:
Overall Officials: Brian Levine, PhD, Principal Investigator — Baycrest Health Sciences
Locations (1):
- Baycrest Health Sciences, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Burgess PW, Alderman N, Evans J, Emslie H, Wilson BA. The ecological validity of tests of executive function. J Int Neuropsychol Soc. 1998 Nov;4(6):547-58. doi: 10.1017/s1355617798466037. PMID 10050359
- [Background] Broadbent DE, Cooper PF, FitzGerald P, Parkes KR. The Cognitive Failures Questionnaire (CFQ) and its correlates. Br J Clin Psychol. 1982 Feb;21(1):1-16. doi: 10.1111/j.2044-8260.1982.tb01421.x. PMID 7126941
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Levine B, Robertson IH, Clare L, Carter G, Hong J, Wilson BA, Duncan J, Stuss DT. Rehabilitation of executive functioning: an experimental-clinical validation of goal management training. J Int Neuropsychol Soc. 2000 Mar;6(3):299-312. doi: 10.1017/s1355617700633052. PMID 10824502
- [Background] Levine B, Schweizer TA, O'Connor C, Turner G, Gillingham S, Stuss DT, Manly T, Robertson IH. Rehabilitation of executive functioning in patients with frontal lobe brain damage with goal management training. Front Hum Neurosci. 2011 Feb 17;5:9. doi: 10.3389/fnhum.2011.00009. eCollection 2011. PMID 21369362
- [Background] Levine B, Stuss DT, Winocur G, Binns MA, Fahy L, Mandic M, Bridges K, Robertson IH. Cognitive rehabilitation in the elderly: effects on strategic behavior in relation to goal management. J Int Neuropsychol Soc. 2007 Jan;13(1):143-52. doi: 10.1017/S1355617707070178. PMID 17166313
- [Background] Hampshire A, Highfield RR, Parkin BL, Owen AM. Fractionating human intelligence. Neuron. 2012 Dec 20;76(6):1225-37. doi: 10.1016/j.neuron.2012.06.022. PMID 23259956
- [Background] Troyer AK, Murphy KJ, Anderson ND, Craik FI, Moscovitch M, Maione A, Gao F. Associative recognition in mild cognitive impairment: relationship to hippocampal volume and apolipoprotein E. Neuropsychologia. 2012 Dec;50(14):3721-8. doi: 10.1016/j.neuropsychologia.2012.10.018. Epub 2012 Oct 24. PMID 23103838
- [Background] Stamenova V, Levine B. Effectiveness of goal management training(R) in improving executive functions: A meta-analysis. Neuropsychol Rehabil. 2019 Dec;29(10):1569-1599. doi: 10.1080/09602011.2018.1438294. Epub 2018 Mar 14. PMID 29540124